CLINICAL TRIAL: NCT05147974
Title: Evaluating the Effectiveness of a Self-management Transdiagnostic Cognitive, Behavioral, Circadian Treatment on Patient Centered Outcomes Such as Self-efficacy, Pain Control and Overall Quality of Life in the Young Adult Chronic Pain Population
Brief Title: The Young Adult Clinic (YAC) Study
Acronym: YAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0075-B
Record Dates: First submitted 2021-11-26; First posted 2021-12-07 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Insomnia; Chronic Pain; Insomnia Due to Medical Condition
Keywords: Insomnia; Pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain; Pain

STUDY DESIGN:
Intervention Model Description: This is a clinical trial as the DOZE app intervention is being assessed for improving outcomes in the YAC patient population.
  We propose a cohort of the YAC patients to be studied, pre & post-intervention, prospectively.
  All participants will be assigned to the intervention (complete DOZE app: Sleep diary and DOZE modules).
  Optional Actigraphy device use for measuring physical activity, sedentary behavior, sleep health parameters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): A cohort of YAC patients to be studied, pre & post-intervention, prospectively. All participants will be assigned to the intervention (complete DOZE app: Sleep diary and DOZE modules).
  Interventions: Behavioral: DOZE app

INTERVENTIONS:
Behavioral: DOZE app — Complete DOZE app: Delivering Online "ZZZ's with Empirical support (DOZE) app plus a Consensus Sleep Diary (CSD).
  The DOZE app, is a web-based app optimized for desktop, smartphone, or tablet use. It is a self-management program for adolescents and young adults with sleep problems. The intervention will be delivered on restricted password-protected applications that will allow tracking of adherence (number of logins to app and website using Google Analytics). Participants will be encouraged to log onto the sleep dairy (via automated alerts) once a day over a 10-week period to complete sleep diary entries, develop and track their goals, and receive sleep health education/tailored sleep health interventions.
  1-week pre- and post- intervention, participants will complete a battery of baseline study questionnaires and have the option of using a Geneactiv actigraphy device along with a CSD.

SUMMARY:
The overarching aim of the Young Adult Clinic (YAC) study is to evaluate the DOZE app, a digital, transdiagnostic behavioral sleep medicine and self-management approach in young adult patients (ages 18-25) with chronic pain.

DETAILED DESCRIPTION:
Sleep, activity, and pain interactions have the potential to impact almost all important protective and regulatory processes in the body. Long-term sleep disruption is associated with increased pain sensitivity, prolonged pain duration, and development of chronic pain. Degree of pain relief can directly impact the quality and disruption of sleep, mood, behavior, social participation, and has a devastating impact on Health Related Quality of Life (HRQL).

Transdiagnostic behavioral sleep medicine and self-management is a behavioral modification approach and is currently a frontline therapy like Cognitive behavioral therapy for insomnia (CBTi) in adults with sleep disorders. However, it is still in early stages of development for adolescent and young adult populations, and less so for youth with co-morbid mental and physical health conditions and chronic pain.

Primary aim: Assess the feasibility of implementing the DOZE app.

Secondary aim:

1. To examine the variance in effectiveness outcomes, including sleep health, pain, and overall Health Related Quality of Life (HRQL).
2. To determine the required sample size for a future definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Young adult patients aged 18 - 25 years old, who have
* Non-malignant chronic pain lasting more than 3 months, with
* Clinically assessed as having a sleep disorder
* English speaking with
* Access to a mobile phone or a computer with internet access.

Exclusion Criteria:

* Patients who require urgent CBT treatment as per their health care provider
* Patients who have received CBT in the past 3 months
* Patients participating in other psychological treatments and/or drug trials during the study
* Patients who have other significant medical conditions- Life threatening (e.g. cancer), neurological conditions (e.g. epilepsy)
* Patients who have other significant psychiatric conditions-Severe depression or active suicide intent
* Situations resulting in forced sleep disruption or derangement of sleep schedule such as night shift work > 2 nights per week in the past 3months
* Pregnancy or breastfeeding.
* Inability to communicate with health care providers or the research personnel
* Inability to fill out self-report questionnaires, study materials, or follow instructions.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Study recruitment/retention | 12 weeks
  Number of Participants recruited/dropping out of study (accrual/dropout rates)
Study compliance to DOZE app intervention/Sleep diary | 10 weeks
  Number of Participants completing/using the DOZE app and completing the sleep diary daily during 10 weeks study intervention
Study DOZE app treatment evaluation | 12 weeks
  Participants' scoring on a 5 point Likert scale pre and post study intervention
Issues and concerns reported via phone calls and emails (Fidelity) | 12 weeks
  Issues and concerns reported while using the intervention tracked by a research assistant, control strategy or outcome measures will be monitored. Can the intervention, and outcome measures be completed as planned or patient not comply with use.

SECONDARY OUTCOMES:
Patient reported improvement in pain | 12 weeks
  Number of Participants reporting Pain Inventory on a brief pain inventory scale of 0 to10.
Patient reported improvement in Health Related Quality Of Life | 12 weeks
  Assessment of pain disability and intensity.PROMIS-29 A 29 item Questionnaire to assets physical, mental and social health and wellbeing.
Patient reported Global Impression of Change | 12 weeks
  Number of Participants reporting an improvement in PGIC in Questionnaire. It comprises 2 scales: PGIC has a 7-point scale depicting a patient's rating of overall improvement (from 1- worse/no change to 7- greatly better/considerable improvement; and a 10-point likert scale rating of efficacy of treatment (where 0- is much better and 10- is much worse).
Patient reported improvement in sleep | 12 weeks
  Adolescent sleep hygiene scale- 28 item self reported questionnaire Never (0%) Once in a while (20%) Sometimes (40%) Quite often (60%) Frequently, but not always (80%) Always (100%)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, M.D, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No